CLINICAL TRIAL: NCT02741050
Title: Camino a La Salud: Adapting and Testing a Primary Care-Delivered Physical Activity Intervention for Latinas With Type II Diabetes
Brief Title: Primary Care-Based Physical Activity for Diabetic Latinas
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: poor recruitment & retention
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Britta Larsen, Assistant Professor, Department of Family Medicine and Public Health, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: K01DK101650 (NIH)
Record Dates: First submitted 2016-04-05; First posted 2016-04-18 (Estimated); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Diabetes; Sedentary Lifestyle
MeSH Terms: conditions — Diabetes Mellitus; Sedentary Behavior | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tailored Physical Activity Intervention (Experimental): Intervention group will receive Spanish-language physical activity print intervention based on SCT and Transtheoretical Model, (TTM) that emphasizes behavioral strategies for increasing activity levels.
  Interventions: Behavioral: Tailored Physical Activity Intervention
- Standard of Care Control Group (Active Comparator): Control group will receive standard of care through the Family Medicine clinic as well as monthly questionnaires on topics other than physical activity (e.g. diet) to complete.
  Interventions: Behavioral: Standard of Care

INTERVENTIONS:
Behavioral: Tailored Physical Activity Intervention — The Tailored Internet intervention is based on constructs of the Transtheoretical Model (TTM) and Social Cognitive Theory (SCT). During the 6-month intervention period, participants will receive monthly mailed questionnaires that assess current motivational readiness for physical activity and other TTM and SCT constructs (e.g., process of change, self-efficacy) and monthly logs to record their current activity.
  Other Names: Camino a La Salud
  Arms: Tailored Physical Activity Intervention
Behavioral: Standard of Care — Those assigned to the control group will continue to receive standard of care through the Family Medicine clinic. This currently entails commonly accepted medication treatment strategies, educational materials and counseling for self-management and medication adherence, screening for depression or other conditions that would impair self-management, and national and state quality of care guidelines for lab testing and control targets (HbA1c, lipids, blood pressure). Participants in the control group will also receive monthly questionnaires on topics other than physical activity (e.g. diet) to fill out and return in order to have the same opportunities for compensation as those in the intervention condition.
  Arms: Standard of Care Control Group

SUMMARY:
The goal of this proposal is to test the efficacy of a primary care-delivered, print-based physical activity intervention for Latinas with type II diabetes. The investigators will test the efficacy of this intervention by randomizing 80 Latinas with type II diabetes recruited through UCSD Health System primary care to either the adapted web-based physical activity intervention or standard of care, and assessing physical activity gains at six and 12 months. The ultimate goal is to develop a print-based physical activity intervention for diabetic Latinas that could be widely disseminated through primary care.

DETAILED DESCRIPTION:
Studies show that adoption of regular physical activity (PA) can greatly enhance diabetes management and prevention. Individuals who adopt a PA routine show significant improvements in clinical markers of diabetes, including HbA1c, glucose tolerance, insulin sensitivity, weight and waist circumference, and significant reductions in medication use, and also show reductions in cardiovascular risk factors and other related co-morbidities. Incorporation of cost-effective PA interventions into primary care for diabetes treatment could therefore enhance overall health and quality of life and significantly reduce healthcare costs. The primary aim of this study is to conduct a small randomized trial (N=80) to test the efficacy of an individually tailored culturally adapted print-based physical activity intervention integrated into primary care to increase weekly moderate-to-vigorous physical activity in Latinas with type II diabetes, compared to those receiving standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Have received a physician's diagnosis of type II diabetes and are currently being seen by a primary care physician
* Currently inactive, defined as participating in at least moderate intensity physical activity for less than 60 minutes per week

Exclusion Criteria:

* Medical condition that may make exercise unsafe, including congestive heart failure, severe musculoskeletal problems or pulmonary conditions, or other conditions determined by the referring physician to preclude unsupervised exercise
* Unable to receive mailed materials (do not have a mailing address)
* Unable to engage in physical activity for at least 30 minutes
* Have a current or planned pregnancy
* Planning to move from the area within the next year

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2019-10 (Actual); Study Completion 2019-10 (Actual)

PRIMARY OUTCOMES:
Objective Changes in Physical Activity from Baseline to 6 Months | Baseline, 6 Months (MO)
  The ActiGraph GT3X+ accelerometer will be the primary measure to assess objective changes in physical activity from baseline to 6 months.
Self-Report Changes in Physical Activity from Baseline to 6 Months | Baseline, 6 Months (MO)
  The 7-Day Physical Activity Recall (PAR) will also assess self-reported changes in physical activity from baseline to 6 months. The 7-Day PAR is an interviewer administered instrument that uses multiple strategies for increasing accuracy of participant recall regarding many types of activities such as time spent sleeping and moderate, hard, and very hard intensity activities. The 7-Day PAR is used across many studies assessing physical activity and has consistently demonstrated acceptable reliability, internal consistency, and congruent validity with other objective measures of activity levels.

SECONDARY OUTCOMES:
Objective Changes in Physical Activity from 6 Months to 12 Months | 6 Months (MO), 12 Months (MO)
  The ActiGraph GT3X+ accelerometer will be the primary measure to assess objective changes in physical activity from 6 to 12 months.
Self-Report Changes in Physical Activity from 6 Months to 12 Months | 6 Months (MO), 12 Months (MO)
  The 7-Day Physical Activity Recall (PAR) will also assess self-reported changes in physical activity from 6 to 12 months. The 7-Day PAR is an interviewer administered instrument that uses multiple strategies for increasing accuracy of participant recall regarding many types of activities such as time spent sleeping and moderate, hard, and very hard intensity activities. The 7-Day PAR is used across many studies assessing physical activity and has consistently demonstrated acceptable reliability, internal consistency, and congruent validity with other objective measures of activity levels.

CONTACTS AND LOCATIONS:
Overall Officials: Britta Larsen, PhD, Principal Investigator — UC, San Diego Department of Family Medicine and Public Health
Locations (1):
- University of California, San Diego, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No